CLINICAL TRIAL: NCT00270348
Title: A Phase III, Multicenter, Double-Blind, Placebo Controlled, Non-Inferiority Study Assessing the Effects of Ciclesonide Metered Dose Inhaler 50 Mg/Day and 200 Mg/Day (Ex-Valve) Administered Once Daily on Growth in Children With Mild Persistent Asthma
Brief Title: Effects of Ciclesonide MDI 50mg/Day and 200mg/Day (Ex-Valve) Once-Daily on Growth in Children With Mild Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTS6159; XRP1526B - 343
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2005-12-28 (Estimated); Status verified 2005-12

CONDITIONS: Asthma
Keywords: Asthma; Safety; Pediatrics
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: ciclesonide

SUMMARY:
The primary objective is to determine if CIC 50 mg/day or 200 mg/day (ex-valve) administered once daily in the morning is non-inferior to placebo with respect to growth velocity in children with mild persistent asthma following a 12-month treatment period

The secondary objective is to investigate changes in growth in terms of bone age (wrist X-ray), and maintenance of asthma control and safety with ciclesonide

ELIGIBILITY:
Inclusion Criteria:

* Females between 5 and 7.5 years and male between 5 and 8.5 years of age with normal heights, a history of mild persistent asthma for at least 3 months prior to visit 1, a forced expiratory volume in one second (FEV1) of ³80% of predicted following at least a 4-hour albuterol withhold, and treated with non-corticosteroid asthma medications on an as-needed or daily basis, or with low doses of inhaled corticosteroids (ICSs) for at least one month prior to Visit 1. Subjects were to be no greater than Stage 1 in the Tanner classification of sexual maturity, and they had to be able to demonstrate effective use of the MDI devices and perform reproducible pulmonary function test.

Exclusion Criteria:

* Subjects with a history of life-threatening asthma, severe respiratory impairment, history of abnormal growth, concurrent disease or condition which may substantially affect growth, previous requirement for daily or alternate day oral corticosteroids (OCS) treatment for ³60 days within the 2 years of Visit 3 and/or any use of OCS within 30 days prior to Visit 1 or during the run-in period, previous treatment with moderate or high doses of inhaled corticosteroid during the 30 days prior to Visit 1

Ages: 5 Years to 102 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450
Dates: Start 2000-12; Study Completion 2004-09

PRIMARY OUTCOMES:
Subject's height measured w. standard stadiometry techniques. 4 acceptable serial measurements taken at each visit on same equipment by a qualified technician.Median of 4 measurements used the subject's stadiometer height data

SECONDARY OUTCOMES:
Blinded assessment of bone age according to Greulich and Pyle radiographic atlas with wrist X-rays. Subjects monitored for AEs and any events occurring during study. Pulmonary function tests performed to measure FEV1 in liters and % of predicted FEV1

REFERENCES:
- [Derived] Skoner DP, Maspero J, Banerji D; Ciclesonide Pediatric Growth Study Group. Assessment of the long-term safety of inhaled ciclesonide on growth in children with asthma. Pediatrics. 2008 Jan;121(1):e1-14. doi: 10.1542/peds.2006-2206. Epub 2007 Dec 10. PMID 18070931